CLINICAL TRIAL: NCT05679830
Title: A Randomized, Open-Label Trial on the Effects of Cannabidiol Isolate on Menstrual-Related Symptoms
Brief Title: The Effects of CBD Isolate on Menstrual-Related Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canopy Growth Corporation (Industry)
Collaborators: James Madison University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRS
Record Dates: First submitted 2022-12-24; First posted 2023-01-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2022-12

CONDITIONS: Menstrual Discomfort
Keywords: cannabidiol; CBD; menstruation
MeSH Terms: interventions — Cannabidiol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 160mg Cannabidiol Isolate (Experimental): 320mg of CBD Isolate BID for 5 days every month starting the day that participants believed they were having menstrual-related symptoms (MRS).
  Interventions: Drug: Cannabidiol
- 320mg Cannabidiol Isolate (Experimental): 160mg of CBD Isolate BID for 5 days every month starting the day that participants believed they were having menstrual-related symptoms (MRS).
  Interventions: Drug: Cannabidiol

INTERVENTIONS:
Drug: Cannabidiol — Cannabidiol is a non-psychoactive cannabinoid obtained from the cannabis plant.

SUMMARY:
The goal of this open-label clinical trial is to compared two different doses for treating menstrual-related symptoms in individuals who experience regular menstrual cycles (occurring for 4-8 days every 21-28 days). The main question it aims to answer is:

(1) if there are changes in menstrual-related symptoms from baseline compared to all 3-months of cannabidiol (CBD) isolate consumption.

Participants will complete a monthly baseline measure after they stop menstruating followed by taking CBD twice daily (BID) for five days for three menstrual cycles and complete the same measures. Researchers will compare 160mg of daily CBD isolate to 320mg of CBD isolate to see if there are differential effects on menstrual-related symptoms (MRS).

ELIGIBILITY:
Inclusion Criteria:

1. Participant is at least 18 years old.
2. Participant is willing and able to provide informed consent and participate in the study for 4 months.
3. Participant experiences a regular period (occurring every 21-38 days and lasting between 4-8 days).
4. Participant is diagnosed with Pre-menstrual Dysphoric Disorder or scores at least '30' on the Menstrual-Related Symptom Questionnaire
5. Participant is willing to begin tracking their periods and menstrual symptoms for the duration of the study
6. Participant agrees to abide by all study restrictions and comply with all study procedures.

Exclusion Criteria:

1. Participant has a known history of significant allergic condition, significant hypersensitivity to CBD, or allergic reaction to cannabis, cannabinoid medications, or excipients of the drug product.
2. Participant has been exposed to any investigational drug or device < 30 days prior to screening or plans to take another investigational drug at any time during the study.
3. Participant has self-reported using cannabis, synthetic cannabinoid or cannabinoid analogue (e.g., dronabinol, nabilone), synthetic cannabinoid receptor agonist (e.g., spice, K2), or any CBD or Tetrahydrocannabinol (THC)-containing product within 30 days of screening or during the study.
4. Participant has a current or past primary Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 diagnosis that the Investigator(s) determines would interfere in treatment or interfere in evaluation of the study treatment (e.g., current psychotic disorder).
5. Participant is currently prescribed medications with known THC- or CBD- interactions (e.g., warfarin, clobazam, valproic acid, phenobarbital, Mammalian target of rapamycin (mTOR) inhibitors, oral tacrolimus).
6. Participant is trying to get pregnant.
7. Participant is pregnant.
8. Participant has a history of suicide attempt in the last year.
9. Participant endorses current suicidal plan and intent during screening.
10. Any other significant disease or disorder which, in the opinion of the investigator, may either put the student at risk because of participation in the study, may influence the result of the study, or affect the student's ability to participate in the study.
11. Participant has a BMI of underweight (18 kg/m2 and below) or obese (30 kg/m2 and above).

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2021-09-23 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Menstrual-Related Symptoms Questionnaire (MRSQ) | 1 menstrual cycle/1 month
  Change in menstrual-related symptoms from baseline scores as measured by the MRSQ every cycle for three cycles. Scores range from 26-104, with higher scores representing greater severity of symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica G Irons, PhD, Principal Investigator — James Madison University
Locations (1):
- James Madison University, Harrisonburg, Virginia, United States